CLINICAL TRIAL: NCT04105998
Title: Effects of Intramuscular Oxytocin on Pupil Diameter and Heart Rate Variability
Brief Title: Effects of Intramuscular (IM) Oxytocin on Pupil Diameter and Heart Rate Variability (HRV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00060838
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2021-11

CONDITIONS: Chronic Pain Due to Injury
Keywords: Healthy Volunteer; Oxytocin; Pupillometry
MeSH Terms: interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blinded crossover treatment with oxytocin and placebo (saline)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, and outcomes assessor will be blinded. The Research Pharmacist will prepare the study medication and hold the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin First, then Placebo (Experimental): Subjects in this arm will receive Intramuscular injection of Oxytocin (Pitocin®), 10 International Units (IU) at the first visit. Then at the next visit, they will receive Intramuscular injection of (1 milliliter) saline.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo, Then Oxytocin (Experimental): Subjects in this arm will receive intramuscular injection of (1 milliliter) saline at the first visit. Then at the next visit, they will receive Intramuscular injection of Oxytocin (Pitocin®), 10 International Units (IU).
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10 IU
  Other Names: Pitocin
Drug: Placebo — Placebo
  Other Names: saline

SUMMARY:
The goal of this study is to test the effects of oxytocin on heart rate variability and pupil diameter, both of which have subtle effects on the activity rate of the autonomic nervous system.

DETAILED DESCRIPTION:
This protocol focuses on two measures of autonomic control to quantify central actions of oxytocin. First, the study team proposes to examine the influence of oxytocin on heart rate variability with focus on its effect on high frequency variability, most commonly ascribed to parasympathetic nervous system activity acting to brake sympathetic tone. Intranasal oxytocin has been demonstrated to have a large effect size on this measure which can be repeated at frequent intervals. As a secondary assessment of parasympathetic activity, the study team will measure low frequency fluctuation in pupil diameter, termed hippus, which also reflects parasympathetic nervous system activity. This outcome measure can be assessed in 3 seconds using equipment currently being used under Institutional Review Board (IRB) approved protocols.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and < 66 years of age,
* Body Mass Index (BMI) <40
* Generally in good health as determined by the Principal Investigator based on prior medical history
* Normal blood pressure and resting heart rate without medication

Exclusion Criteria:

* Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk
* Women who are pregnant (positive result for serum pregnancy test at screening visit),
* Women who are currently nursing or lactating, women that have been pregnant within 2 years.
* Neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
* Previous eye surgery, eye medications, cataracts

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norman GJ, Cacioppo JT, Morris JS, Malarkey WB, Berntson GG, Devries AC. Oxytocin increases autonomic cardiac control: moderation by loneliness. Biol Psychol. 2011 Mar;86(3):174-80. doi: 10.1016/j.biopsycho.2010.11.006. Epub 2010 Nov 30. PMID 21126557
- [Background] Turnbull PR, Irani N, Lim N, Phillips JR. Origins of Pupillary Hippus in the Autonomic Nervous System. Invest Ophthalmol Vis Sci. 2017 Jan 1;58(1):197-203. doi: 10.1167/iovs.16-20785. PMID 28114580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed via advertising in the community and internally within the medical center. Subjects who met inclusion criteria were scheduled for a visit at the Pain Research Clinical Research Unit where the written informed consent was obtained. The enrollment period was 10/24/2019 to 11/01/2021
Groups:
- Oxytocin First: Participant received intravenous oxytocin, 10 IU on study day 1 and placebo on study day 2
- Placebo First: Participant received intravenous placebo on study day 1 and oxytocin, 10 IU on study day 2
Period: First Study Day
Arm/Group | Oxytocin First | Placebo First
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0
Period: Second Study Day
Arm/Group | Oxytocin First | Placebo First
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Altered frequency and times of measurements on both study days | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin on Study Day 1 and Placebo Study Day 2: Participant received intravenous oxytocin, 10 International Units (IU) on study day 1 and intravenous placebo on study day 2
- Placebo on Study Day 1 and Placebo: Participant received intravenous placebo on study day 1 and intravenous oxytocin, 10 International Units (IU) on study day 2
- Total: Total of all reporting groups
Arm/Group | Oxytocin on Study Day 1 and Placebo Study Day 2 | Placebo on Study Day 1 and Placebo | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12) | 35 (15) | 35 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Fluctuation in Pupil Diameter (Hippus) -Pre Drug Administration
Description: Magnitude of power at the dominant frequency in the Fourier transform of pupil diameter in the .1-2 Hz range, termed hippus. Pupil measurements will be made for 20 seconds every 5 minutes for 20 minutes. The Fast Fourier Transform (FFT) essentially takes what looks like a random, noisy signal and distills it into a combination of many sine waves, each with different frequencies and different sizes (think ocean waves, which has the big wave we see and the small up and down wavelets on the top of the water). The primary outcome measure is the size of the largest wave in the frequency range above in this FFT analysis. Its dimensions are milliseconds^2.
Time Frame: From 20 minutes before until study drug injection
Measure: Mean (Standard Deviation); unit: milliseconds^2
Groups:
- Oxytocin: Participant received intravenous oxytocin, 10 International Units (IU) on study day 1 or 2
- Placebo: Participant received intravenous placebo on study day 1 or 2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 20 | 20
milliseconds^2 | 1.61 (1.20) | 1.71 (1.26)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.64, t-test, 2 sided

2. Primary Outcome: Fluctuation in Pupil Diameter (Hippus) -Post Drug Administration
Description: Magnitude of power at the dominant frequency in the Fourier transform of pupil diameter in the .1-2 Hz range, termed hippus. Pupil measurements will be made for 20 seconds every 5 minutes until 90 minutes after study drug administration. The Fast Fourier Transform (FFT) essentially takes what looks like a random, noisy signal and distills it into a combination of many sine waves, each with different frequencies and different sizes (think ocean waves, which has the big wave we see and the small up and down wavelets on the top of the water). The primary outcome measure is the size of the largest wave in the frequency range above in this FFT analysis. Its dimensions are milliseconds^2.
Time Frame: For 90 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 20 | 20
milliseconds^2 | 1.34 (0.56) | 1.52 (0.68)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.19, t-test, 2 sided

3. Primary Outcome: Fluctuation in Pupil Diameter (Hippus) -Post Drug Administration
Description: Magnitude of power at the dominant frequency in the Fourier transform of pupil diameter in the .1-2 Hz range, termed hippus. Pupil measurements will be made for 20 seconds every 5 minutes until 120 minutes after study drug administration. The Fast Fourier Transform (FFT) essentially takes what looks like a random, noisy signal and distills it into a combination of many sine waves, each with different frequencies and different sizes (think ocean waves, which has the big wave we see and the small up and down wavelets on the top of the water). The primary outcome measure is the size of the largest wave in the frequency range above in this FFT analysis. Its dimensions are milliseconds^2.
Time Frame: For 120 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 7 | 7
milliseconds^2 | 0.98 (0.54) | 1.49 (1.39)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.067, t-test, 2 sided

4. Primary Outcome: Heart Rate Variability in the High Frequency Range
Description: Magnitude of peak power in the 0.12-0.40 Hz frequency range of the Fast Fourier Transform of heart rate. The Fast Fourier Transform (FFT) essentially takes what looks like a random, noisy signal and distills it into a combination of many sine waves, each with different frequencies and different sizes (think ocean waves, which has the big wave we see and the small up and down wavelets on the top of the water). The primary outcome measure is the size of the largest wave in the frequency range above in this FFT analysis. Its dimensions are milliseconds^2.
Time Frame: From 20 minutes before until study drug injection
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 20 | 20
milliseconds^2 | 182 (151) | 253 (296)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.25, t-test, 2 sided

5. Primary Outcome: Heart Rate Variability in the High Frequency Range
Description: as for outcome 4
Time Frame: For 90 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 20 | 20
milliseconds^2 | 183 (158) | 300 (296)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.058, t-test, 2 sided

6. Primary Outcome: Heart Rate Variability in the High Frequency Range
Description: as for outcome 4
Time Frame: For 120 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 7 | 7
milliseconds^2 | 247 (216) | 381 (273)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.111, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 days
Description: Participants were asked to describe any adverse events that have been reported after oxytocin administration, including headache, facial flushing, sensation of heart pounding, or abdominal or pelvic cramping during and for one hour after infusion of study drug. They were contacted at 1 and 7 days after study drug administration and queried for these or other adverse events.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04105998/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT04105998/ICF_000.pdf